CLINICAL TRIAL: NCT02965963
Title: The Effect of Dopamine on Pulmonary Diffusion and Capillary Blood Volume During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00067664
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Health
MeSH Terms: interventions — Dopamine; Metoclopramide; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Dopamine (Experimental): Dependent variables measured with intravenous low dose dopamine infusion at rest, 60%, and 85% of VO2max
  Interventions: Drug: Dopamine; Other: Rest; Other: Exercise - 60%; Other: Exercise - 85%
- Metoclopramide (Experimental): Dependent variables measured with oral metoclopramide ingestion at rest, 60%, and 85% of VO2max
  Interventions: Drug: Metoclopramide; Other: Rest; Other: Exercise - 60%; Other: Exercise - 85%
- Placebos (Experimental): Dependent variables measured with orally ingested placebo pill and intravenous saline at rest, 60%, and 85% of VO2max
  Interventions: Drug: Placebos; Other: Rest; Other: Exercise - 60%; Other: Exercise - 85%

INTERVENTIONS:
Drug: Dopamine
  Arms: Dopamine
Drug: Metoclopramide
  Arms: Metoclopramide
Drug: Placebos
  Arms: Placebos
Other: Rest
Other: Exercise - 60% — 60% of VO2max
Other: Exercise - 85% — 85% of VO2max

SUMMARY:
The purpose of this study is to examine the effect of dopamine infusion and dopamine-2 receptor blockade on pulmonary capillary blood volume, diffusion, and the hemodynamic variables of pulmonary artery pressure, cardiac output, and pulmonary vascular resistance during exercise. Secondarily, this study will examine the effect of dopamine infusion and dopamine-2 receptor blockade on exercise tolerance.

DETAILED DESCRIPTION:
1. Study Objectives

   The primary objective of this study is to examine the effect of dopamine infusion and dopamine-2 receptor blockade on pulmonary capillary blood volume, diffusion, and the hemodynamic variables of pulmonary artery pressure, cardiac output, and pulmonary vascular resistance during exercise. Secondarily, this study will examine the effect of dopamine infusion and dopamine-2 receptor blockade on exercise tolerance.
2. Background

   To meet the increased oxygen demand required for exercise, pulmonary diffusing capacity (DLCO) must increase in order to avoid a drop in arterial oxygenation and early exercise termination. Enhanced DLCO during exercise is achieved by expanding pulmonary capillary blood volume (Vc) and diffusing membrane capacity (Dm) through recruitment and distention of the pulmonary capillaries, effectively increasing the surface area for diffusion. Recruitment and distention of the pulmonary capillaries decreases pulmonary vascular resistance (PVR), increasing pulmonary blood flow (Q) while limiting the rise in pulmonary artery pressure (PAP) with exercise.

   In health, pharmacological interventions are not believed to affect PAP during exercise. However, dopamine, a pulmonary vasodilator, may help to regulate PAP during exercise. Specifically, dopamine appears important for a normal cardiovascular exercise response, as Metoclopramide (pulmonary dopamine-2-receptor antagonist) decreases maximal Q and exercise tolerance (1). These results suggest that dopamine may modulate Vc during exercise via pulmonary smooth muscle regulation, subsequently affecting PVR, PAP, Q and exercise tolerance. However, how dopamine regulates DLCO, Vc, Q, and exercise tolerance is unknown.

   Purpose: The purpose of this study is to examine the effect of a dopamine agonist and a dopamine-2-receptor antagonist on DLCO, Vc, PAP, PVR, Q, and exercise tolerance.

   Hypothesis: It is hypothesized that dopamine will increase Vc, leading to a reduction in PVR and a corresponding decrease in PAP. This response will allow an increase in DLCO, Q, and exercise tolerance relative to control. Conversely, Metoclopramide (dopamine-2-receptor antagonist) will attenuate the increase in Vc as well as the reduction in PVR, leading to an increase in PAP. In this condition, DLCO, Q, and exercise tolerance will be reduced.
3. Methods

Study Overview: This study will utilize a randomized, double-blind crossover design where healthy subjects will have measurements performed at rest and 2 workloads (60% and 85% of previously determined VO2peak) with either intravenous dopamine (2µg/kg/min), dopamine receptor blockade (20mg oral Metoclopramide), or placebo (order randomized). Data will be collected across 5 different days over a 2-3 week period. Day 1: Pulmonary function and graded exercise testing to exhaustion. Day 2-4: Vc determination at rest and exercise with either intravenous dopamine, dopamine receptor blockade, or placebo (order randomized). Following a brief period of rest, time to exhaustion trials at 85% of VO2peak will be performed to characterize exercise tolerance. Day 5: Evaluation of PAP via cardiac ultrasound at rest and during exercise with either intravenous dopamine, dopamine receptor blockade, or placebo (order randomized).

Pulmonary Function & Cardiopulmonary Exercise Test: Subjects will undergo a graded exercise test to volitional exhaustion to characterize aerobic fitness (VO2peak) and a standard pulmonary function test to characterize lung function parameters.

DLCO and Vc measurement during exercise: DLCO and Vc will be measured using the multiple oxygen tension DLCO breath-hold method (2) at rest and during cycling exercise at 60% and 85% of VO2peak. Over different three days, participants will be randomized to each of the following conditions: 1) dopamine (2 μg/kg/min intravenous) and a placebo pill, 2) metoclopramide (20 mg oral) and intravenous saline, or 3) intravenous saline and a placebo pill. During each workload, subjects will perform a DLCO breath-hold maneuver for six seconds, repeated three times during exercise at differing oxygen tensions (0.21, 0.40, 0.60; workload and oxygen tension randomized) allowing for calculation of Vc and Dm. Trials will be spread over several days to ensure no CO buildup. DLCO will be corrected for hemoglobin, and we have considerable experience in performing these tests.

Pulmonary Artery Systolic Pressure (PASP), PVR, and Q: Doppler echocardiography (PASP) will be used as a non-invasive estimate of PAP in all dopamine conditions. PASP will be evaluated at rest and during exercise, and this method has been used successfully by our group and others in previous investigations(3,4). Total PVR will be evaluated by dividing PASP by Q at any given workload. Q will be evaluated using the Physioflow® Impedance Cardiography (Manatec® Biomedical). When compared to direct Fick methods, impedance cardiography provides an accurate determination of Q at rest and during exercise.

Hemoglobin: Since DLCO will be corrected for hemoglobin concentration, a small sample of blood will be collected via finger prick at rest and during exercise and analyzed for hemoglobin concentration using a hand-held Hemoglobin measurement device (HemoCue 201+, HemoCue AB, Angelholm, Sweden).

ELIGIBILITY:
Inclusion Criteria:

* Physically active (exercising >2 times per week)
* BMI < 30kg/m2
* No known cardiac or pulmonary disease

Exclusion Criteria:

* Known cardiac or pulmonary diseases / abnormalities
* Use of medications that could interfere with dopaminergic pathways (i.e. dopaminergic agonists / antagonists, alcohol, central nervous system depressants, and serotonergic drugs)
* BMI > 30kg/m2
* Female subjects must not be pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2025-06 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Capillary Blood Volume | Dopamine (Day 1), Metoclopramide (Day 2), Placebos (Day 3) *order randomized
  Roughton and Forster's Three FIO2 DLCO Method at Rest, 60% of Vo2max, and 85% of Vo2max
Diffusing Capacity for Carbon Monoxide | Dopamine (Day 1), Metoclopramide (Day 2), Placebos (Day 3) *order randomized
  Roughton and Forster's Three FIO2 DLCO Method at Rest, 60% of Vo2max, and 85% of Vo2max
Pulmonary Artery Systolic Pressure | Dopamine (Day 1), Metoclopramide (Day 2), Placebos (Day 3) *order randomized
  Non-invasive estimation using Doppler echocardiography at Rest & 60% of Vo2max
Cardiac Output | Dopamine (Day 1), Metoclopramide (Day 2), Placebos (Day 3) *order randomized
  Non-invasive estimation using trans-thoracic impedance cardiography at rest, 60% of Vo2max, and 85% of Vo2max
Pulmonary Vascular Resistance | Dopamine (Day 1), Metoclopramide (Day 2), Placebos (Day 3) *order randomized
  Calculation

SECONDARY OUTCOMES:
Exercise Tolerance | Dopamine (Day 1), Metoclopramide (Day 2), Placebos (Day 3) *order randomized
  Time-to-exhaustion at 85% of VO2max
Exertional Dyspnea | Dopamine (Day 1), Metoclopramide (Day 2), Placebos (Day 3) *order randomized
  Modified Borg scale for Dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Research Laboratory, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Tedjasaputra V, Bryan TL, van Diepen S, Moore LE, Bouwsema MM, Welsh RC, Petersen SR, Stickland MK. Dopamine receptor blockade improves pulmonary gas exchange but decreases exercise performance in healthy humans. J Physiol. 2015 Jul 15;593(14):3147-57. doi: 10.1113/JP270238. Epub 2015 Jun 8. PMID 25952760
- [Background] ROUGHTON FJ, FORSTER RE. Relative importance of diffusion and chemical reaction rates in determining rate of exchange of gases in the human lung, with special reference to true diffusing capacity of pulmonary membrane and volume of blood in the lung capillaries. J Appl Physiol. 1957 Sep;11(2):290-302. doi: 10.1152/jappl.1957.11.2.290. No abstract available. PMID 13475180
- [Background] Argiento P, Chesler N, Mule M, D'Alto M, Bossone E, Unger P, Naeije R. Exercise stress echocardiography for the study of the pulmonary circulation. Eur Respir J. 2010 Jun;35(6):1273-8. doi: 10.1183/09031936.00076009. Epub 2009 Nov 19. PMID 19926746
- [Background] Bryan TL, van Diepen S, Bhutani M, Shanks M, Welsh RC, Stickland MK. The effects of dobutamine and dopamine on intrapulmonary shunt and gas exchange in healthy humans. J Appl Physiol (1985). 2012 Aug 15;113(4):541-8. doi: 10.1152/japplphysiol.00404.2012. Epub 2012 Jun 14. PMID 22700799